CLINICAL TRIAL: NCT05090423
Title: The Effect of Additional Neurodynamic Intervention in Patients With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM110112F
Record Dates: First submitted 2021-09-27; First posted 2021-10-22 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Ankle Sprains
Keywords: Chronic ankle instability; Neurodynamics; Mechanosensitivity
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: balance training alone (Experimental): The subjects will receive 12 sessions of balance training over six to eight weeks.
  Interventions: Other: balance training alone
- Experimental: balance training and neurodynamic intervention for the common peroneal nerve (Experimental): The subjects will receive the 12 sessions of balance training and neurodynamic intervention for the common peroneal nerve over six to eight weeks.
  Interventions: Other: balance training and neurodynamic intervention for the common peroneal nerve

INTERVENTIONS:
Other: balance training alone — The subjects will warm up to stretch the lower extremity for 5 minutes.
  The physical therapist will instruct the patient how to use the foot tripod within 5 minutes. And then, giving him or her balance training.
  At the first, the patient double legs stand on the ground to throw and catch a ball for 30 seconds, and then one leg stand on the ground to throw and catch a ball for 30 seconds. When finished, the patient can take 1 minutes rest.
  Second, the patient will finish the prescribed the task stand on different materials, which included the exercise mat, dynair, bosu and foam roller.
  Arms: Experimental: balance training alone
Other: balance training and neurodynamic intervention for the common peroneal nerve — The physical therapist will give the patient neurodynamic intervention for the common peroneal nerve, which is performed slider the nerve 2 seconds.
  The slider technique is repeated 30 seconds for 4 times, each time can be take a rest 1 minutes.
  The physical therapist will instruct the patient how to use the foot tripod within 5 minutes. And then, giving him or her balance training.
  At the first, the patient double legs stand on the ground to throw and catch a ball for 30 seconds, and then one leg stand on the ground to throw and catch a ball for 30 seconds. When finished, the patient can take 1 minutes rest.
  Second, the patient will finish the prescribed the task stand on different materials, which included the exercise mat, dynair, bosu and foam roller.
  Arms: Experimental: balance training and neurodynamic intervention for the common peroneal nerve

SUMMARY:
Approximately 40% of acute ankle sprain would develop into chronic ankle instability (CAI). Chronic ankle instability is characterized by pain, repeated sprains and giving way. Recently, the pathomechanical impairment, sensory-perceptual impairment and motor-behavioral impairment have been documented in the chronic ankle instability model. Previous research revealed that compared to the control subjects, people with CAI had lower pressure pain threshold (PPT). This increased mechanosensitivity of the neural tissues around the ankle might account for pain and dysfunction in people with CAI. Also, the other study indicated that in subjects following ankle inversion sprain there is greater restriction of knee extension on the injured side compared to non-injured side in the slump test with the ankle plantar flexion and inversion, which may suggest the restriction in mobility of the common peroneal tract. However, the effects of neurodynamic intervention, which addresses the mechanosensitivity problems, in people with CAI are still unclear.

Therefore, the aim of the study is to investigate the effect of additional neurodynamic intervention on the ankle range of motion, mechanosensitivity, balance performance and self-reported function.

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is characterized by pain, repeated sprains and giving way. Approximately 40% of acute ankle sprain would develop into chronic ankle instability. Recently, the pathomechanical impairment, sensory-perceptual impairment and motor-behavioral impairment have been documented in the chronic ankle instability model. Previous research revealed that compared to the control subjects, people with CAI had lower pressure pain threshold (PPT). This increased mechanosensitivity of the neural tissues around the ankle might account for pain and dysfunction in people with CAI. Pahor et al., indicated that in subjects following ankle inversion sprain there is greater restriction of knee extension on the injured side compared to non-injured side in the slump test with the ankle plantar flexion and inversion, which may suggest the restriction in mobility of the common peroneal tract. However, the effects of neurodynamic intervention, which addresses the mechanosensitivity problems, in people with CAI are still unclear. Purpose: The aim of the study is to investigate the effects of neurodynamic intervention on the mechanosensitivity, balance performance and self-reported function in patients with CAI. Study design: A randomized controlled trial design. Single-blinded. Methods: Forty subjects between 20-50 with CAI were recruited and randomized into either the exercise only group or the neurodynamic intervention with exercise (neurodynamic) group. The sample size was calculated based on the PPT data of Lorenzo-Sanchez-Aguilera et al's, which requires 20 subjects in each group to reach a statistical power of 0.8. Both groups were receive 12 interventions within 6-8 weeks. The exercise only group performed balance training, while the neurodynamic group received balance training and neurodynamic intervention for the common peroneal nerve. Outcome measures included demographic data, pressure pain threshold, active knee extension range of motion (ROM) of the slump test with ankle plantarflexion and inversion (AKEOST), hamstrings flexibility, ankle range of motion, Y balance test and foot and ankle ability measure (FAAM).

ELIGIBILITY:
Inclusion Criteria:

1. History of at least two ankle sprains in the same leg, of which the first sprain is more than one year
2. Leading to at least one interrupted day of desired physical activity
3. The Cumberland Ankle Instability Tool (CAIT) ≦ 24
4. Slump test in ankle plantar flexion with inversion: positive

Exclusion Criteria:

1. Pregnancy
2. Surgical treatments
3. Previous fractures in either lower extremity
4. Any concomitant lower extremity pathology, for example, vascular disease, osteoarthritis and rheumatoid arthritis
5. Significant pain or injury to the lumbar or cervical spine
6. Regular use of medication: anti-inflammatory drugs, painkiller, steroid or muscle relaxants
7. Previous manual therapy or exercise interventions received on the lower extremity within the previous 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shih Yi-Fen, Ph.D, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming
Locations (1):
- National Yang Ming University, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, participants with chronic ankle instability were recruited from Yang Ming Chiao Tung University and various orthopedic and rehabilitation clinics in Taipei. Potential participants were first contacted to confirm preliminary eligibility. During the initial meeting, the study process and relevant details were explained. Eligibility was further verified based on inclusion and exclusion criteria. Upon confirmation, participants provided informed consent to participate in the study.
Pre-assignment Details: In this study, 59 participants were initially recruited to meet the inclusion criteria. Among them, 36 participants (14 males and 22 females) were confirmed to meet the eligibility requirements. Due to others not meeting inclusion criteria or falling under exclusion criteria.
Groups:
- Exercise Group: The exercise group receives 12 treatment interventions over six to eight weeks, with each session lasting approximately 20 minutes.
  First, 5-minute warm-up and stretching session, followed by foot core exercises and instruction on foot stability movements. The 12 treatment sessions were divided into three stages based on difficulty.
- Neurodynamic Group: The exercise group underwent 12 treatment sessions over a period of six to eight weeks, each lasting about 20 minutes. Initially, the treatment involved peroneal nerve sliding techniques: movements were executed every two seconds for 30 seconds, repeated four times. Between each session, there was a one-minute rest, totaling five minutes. The 12 sessions of neurodynamic interventions were categorized into three progressive stages. Following this, participants engaged in foot core exercises and received instructions on foot stability movements, also organized into three stages based on difficulty.
Period: Overall Study
Arm/Group | Exercise Group | Neurodynamic Group
Started | 18 | 18
Completed | 15 | 15
Not Completed | 3 | 3
Not completed — Because of the covid-19 | 3 | 2
Not completed — repeated ankle sprain in daily of life | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Neurodynamic Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (4.84) | 25 (4.62) | 24.64 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 18 | 18 | 36
Pressure pain threshold-anterior talofibular ligament [Mean (Standard Deviation); unit: kg/ cm²] — Pressure pain threshold (PPT) was measured using a digital algometer (PainTest™ FDX, Wagner Instruments) applied perpendicularly to the target site. Pressure was increased at a constant rate until the participant first reported pain. Three trials were performed with 30-second intervals between trials. The mean of the three readings was recorded. The unit of measure was kilograms per square centimeter (kg/cm²).
  kg/ cm² | 3.6 (1.29) | 3.38 (0.85) | 3.5 (1.09)
Pressure pain threshold-calcaneofibular ligament [Mean (Standard Deviation); unit: kg/ cm²] | 4.72 (1.37) | 4.14 (0.1) | 4.43 (1.22)
Pressure pain threshold-peroneal brevis muscle [Mean (Standard Deviation); unit: kg/ cm²] | 4.48 (1.41) | 3.73 (1.16) | 4.11 (1.33)
Pressure pain threshold-peroneal longus muscle [Mean (Standard Deviation); unit: kg/ cm²] | 6.39 (1.59) | 5.27 (1.35) | 5.83 (1.56)
Pressure pain threshold-common peroneal nerve [Mean (Standard Deviation); unit: kg/ cm²] | 5.28 (1.49) | 4.21 (1.34) | 4.74 (1.5)
Active knee extension range of motion during slump test in ankle plantar flexion with inversion [Mean (Standard Deviation); unit: degree] | 34.19 (3.39) | 36.39 (3.39) | 35.29 (14.22)
Hamstring flexibility [Mean (Standard Deviation); unit: degree] | 40.63 (2.61) | 41.02 (2.61) | 40.83 (10.93)
Weight-bearing lunge test [Mean (Standard Deviation); unit: degree] — Ankle dorsiflexion was measured using the weight-bearing lunge test (WBLT). Participants performed a forward lunge with the test foot in front. While keeping the heel on the ground, they bent the knee toward the wall. A gravity inclinometer placed on the tibial tuberosity measured the angle between the tibia and floor. After 3 warm-up trials, 3 test trials were recorded and averaged. Unit: degrees (°).
  degree | 44.87 (7.89) | 43.96 (5.36) | 44.42 (6.66)
Y balance test-anterior direction [Mean (Standard Deviation); unit: %] — Dynamic balance was assessed using the Y-Balance Test. Participants stood barefoot on the test foot at the center of the Y-platform, hands on hips, with the toes behind the red line. While keeping the heel down, they used the other foot to reach in anterior, posterolateral, and posteromedial directions without touching the floor or pushing down on the reach indicators. After 6 practice trials, 3 test trials were performed per direction. Reach distances were averaged and normalized to leg length using: (reach distance / leg length) × 100%.
  % | 55.1 (5.28) | 53.05 (5.79) | 54.09 (5.51)
Y balance test-posterolateral direction [Mean (Standard Deviation); unit: %] — Dynamic balance was assessed using the Y-Balance Test. Participants stood barefoot on the test foot at the center of the Y-platform, hands on hips, with the toes behind the red line. While keeping the heel down, they used the other foot to reach in anterior, posterolateral, and posteromedial directions without touching the floor or pushing down on the reach indicators. After 6 practice trials, 3 test trials were performed per direction. Reach distances were averaged and normalized to leg length using: (reach distance / leg length) × 100%.
  % | 94.2 (8.86) | 88.27 (10.75) | 91.22 (10.2)
Y balance test-posteromedial direction [Mean (Standard Deviation); unit: %] — Dynamic balance was assessed using the Y-Balance Test. Participants stood barefoot on the test foot at the center of the Y-platform, hands on hips, with the toes behind the red line. While keeping the heel down, they used the other foot to reach in anterior, posterolateral, and posteromedial directions without touching the floor or pushing down on the reach indicators. After 6 practice trials, 3 test trials were performed per direction. Reach distances were averaged and normalized to leg length using: (reach distance / leg length) × 100%.
  % | 85.09 (7.94) | 84.3 (9.67) | 84.71 (8.7)
Foot and ankle ability measure-Activity of Life [Mean (Standard Deviation); unit: %] — The FAAM includes two subscales: Activities of Daily Living (21 items, max 84 points) and Sports (8 items, max 32 points). Each item is rated from 0 (unable to do) to 4 (no difficulty); N/A responses are excluded. Scores are summed and converted to a percentage. A self-reported global rating (0-100%) is also recorded, where the unaffected foot is considered 100%. Participants completed the form based on activities within the past week.
  % | 92.99 (7.19) | 91.6 (7.81) | 92.29 (7.47)
Foot and ankle ability measure- Activity of Life (Self- Awareness Score) [Mean (Standard Deviation); unit: units on a scale] — The FAAM includes two subscales: Activities of Daily Living (21 items, max 84 points) and Sports (8 items, max 32 points). Each item is rated from 0 (unable to do) to 4 (no difficulty); N/A responses are excluded. Scores are summed and converted to a percentage. A self-reported global rating (0-100%) is also recorded, where the unaffected foot is considered 100%. Participants completed the form based on activities within the past week.
  units on a scale | 84.56 (7.59) | 82.5 (15.46) | 83.53 (12.05)
Foot and ankle ability measure-sports [Mean (Standard Deviation); unit: %] — The FAAM includes two subscales: Activities of Daily Living (21 items, max 84 points) and Sports (8 items, max 32 points). Each item is rated from 0 (unable to do) to 4 (no difficulty); N/A responses are excluded. Scores are summed and converted to a percentage. A self-reported global rating (0-100%) is also recorded, where the unaffected foot is considered 100%. Participants completed the form based on activities within the past week.
  % | 81.15 (13.52) | 81.94 (14.57) | 81.54 (13.81)
Foot and ankle ability measure- Sports (Self- Awareness Score) [Mean (Standard Deviation); unit: units on a scale] — The FAAM includes two subscales: Activities of Daily Living (21 items, max 84 points) and Sports (8 items, max 32 points). Each item is rated from 0 (unable to do) to 4 (no difficulty); N/A responses are excluded. Scores are summed and converted to a percentage. A self-reported global rating (0-100%) is also recorded, where the unaffected foot is considered 100%. Participants completed the form based on activities within the past week.
  units on a scale | 75.56 (11.87) | 72.39 (20) | 73.97 (16.28)

OUTCOME MEASURES:

1. Primary Outcome: Pressure Pain Threshold- Anterior Talofibular Ligament
Description: Using the PainTestTM FDX algometer, apply vertical contact and average force to measure pressure pain thresholds at the anterior talofibular ligament. The point is tested three times with a 30-second interval between tests, and the average of the three measurements is recorded.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: kg/ cm²
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
kg/ cm² | 4.19 (1.3) | 3.98 (1.29)

2. Primary Outcome: Pressure Pain Threshold- Calcaneofibular Ligament
Description: Using the PainTestTM FDX algometer, apply vertical contact and average force to measure pressure pain thresholds at the calcaneofibular ligament. The point is tested three times with a 30-second interval between tests, and the average of the three measurements is recorded.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: kg/ cm²
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
kg/ cm² | 4.98 (1.62) | 4.67 (1.43)

3. Primary Outcome: Active Knee Extension Range of Motion During Slump Test in Ankle Plantar Flexion With Inversion
Description: The subjects sat on the edge of the bed without touching the ground with their feet. The physical therapist assisted the subjects in maintaining a neutral pelvis position. First, the subjects were asked to flex the neck, trunk, and finally the lumbar to tighten the back. Second, while the subjects plantarflexed and inverted the ankle, they performed the knee extension movement, and the angle of knee motion was recorded. Participants performed three practice trials followed by three test trials and averaged the three tests.
Time Frame: Within one week after 12 treatment session
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
degree | 24.53 (1.9) | 17.8 (1.9)
Statistical Analysis 1: Comparison: Exercise Group vs Neurodynamic Group; Test type: Other; p = 0.018, ANOVA

4. Primary Outcome: Pressure Pain Threshold- Peroneal Brevis Muscle
Description: Using the PainTestTM FDX algometer, apply vertical contact and average force to measure pressure pain thresholds at the peroneal brevis muscle. The point is tested three times with a 30-second interval between tests, and the average of the three measurements is recorded.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: kg/ cm²
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
kg/ cm² | 4.66 (1.36) | 4.27 (1.19)

5. Primary Outcome: Pressure Pain Threshold- Peroneal Longus Muscle
Description: Using the PainTestTM FDX algometer, apply vertical contact and average force to measure pressure pain thresholds at the peroneal longus muscle. The point is tested three times with a 30-second interval between tests, and the average of the three measurements is recorded.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: kg/ cm²
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
kg/ cm² | 6.3 (2) | 5.93 (1.5)

6. Primary Outcome: Pressure Pain Threshold- Common Peroneal Nerve
Description: Using the PainTestTM FDX algometer, apply vertical contact and average force to measure pressure pain thresholds at the common peroneal nerve. The point is tested three times with a 30-second interval between tests, and the average of the three measurements is recorded.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: kg/ cm²
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
kg/ cm² | 5.47 (1.58) | 4.89 (1.39)

7. Secondary Outcome: Y Balance Test- Anterior Direction
Description: Participants stood on the Y-Balance Test device and reached with the non-stance leg in the anterior, posterolateral, and posteromedial directions, starting with the dominant leg, in sequence. Each participant performed six practice trials to become familiar with the procedure. For data collection, three final trials in each direction were recorded. Leg length was measured from the anterior superior iliac spine to the distal tip of the medial malleolus. Reach distance in centimeters was normalized to leg length by dividing the reach distance by leg length and multiplying by 100 to obtain the percentage of leg length for statistical analysis.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: % of leg length
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
% of leg length | 61.18 (5.87) | 59.22 (4.01)

8. Secondary Outcome: The Foot and Ankle Ability Measures- Sports
Description: The Foot and Ankle Ability Measure (FAAM) Sports Subscale is a self-reported questionnaire consisting of 8 items that assess the participant's perceived ability to perform sports-related activities. Each item is rated on a 5-point scale (0 = unable to do, 1 = extreme difficulty, 2 = moderate difficulty, 3 = slight difficulty, 4 = no difficulty). If an item is not applicable, the participant marks "N/A."
  Raw scores are summed and converted to a percentage score using the following formula: (raw score ÷ maximum possible score) × 100, with higher scores indicating better functional ability.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
percentage | 93.35 (4.22) | 93.55 (9.58)

9. Secondary Outcome: The Foot and Ankle Ability Measures- Activity of Life
Description: The Foot and Ankle Ability Measure (FAAM) Activities of Daily Living (ADL) subscale is a self-reported questionnaire consisting of 21 items that assess the participant's perceived difficulty in performing activities of daily living. Each item is rated on a 5-point scale (0 = unable to do, 1 = extreme difficulty, 2 = moderate difficulty, 3 = slight difficulty, 4 = no difficulty). If an item is not applicable, the participant marks "N/A."
  Raw scores are summed and converted to a percentage score using the following formula: (raw score ÷ maximum possible score) × 100, with higher scores indicating better functional ability.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
percentage | 98.13 (1.65) | 97.86 (3.32)

10. Secondary Outcome: Weight Bearing Lunge Test
Description: Asked the person to face the wall and placed the tested foot in front, with the second toe and heel in a line perpendicular to the wall. The contralateral limb was positioned behind the testing limb in a comfortable position, and hands were placed on the wall in front to maintain stability. The gravity inclinometer was placed at the tibial tuberosity to measure the angle. The subjects lunged forward, trying to touch a vertical line on the wall with their knee, while keeping their heel in contact with the ground.
  Participants performed three practice trials followed by three test trials and averaged the three tests.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
degree | 41.27 (6.66) | 40.38 (5.09)

11. Secondary Outcome: Hamstring Flexibility
Description: Measured hamstring flexibility using the 90-90 passive knee extension test. The subject lay flat on their back on the bed and straps were used to secure the pelvis. The test leg was positioned with the hip and knee at 90 degrees, while the other leg remained straight on the bed. The subject's knee was then passively extended. The goniometer's stationary arm was attached to the middle of the thigh, the axis was aligned with the lateral epicondyle of the femur, and the moving arm was positioned to the lateral malleolus. The knee extension angle was measured. The value recorded was the angle between the lower leg and the vertical line.
  Participants performed three practice trials followed by three test trials and averaged the three tests.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
degree | 38.07 (2.7) | 30.78 (2.7)

12. Secondary Outcome: The Foot and Ankle Ability Measures- Activity of Life (Self- Awareness Score)
Description: The Activities of Daily Living (self-awareness score) is a self-reported measure in which the participant rates the functional status of the involved (patient) foot relative to the uninvolved (healthy) foot. The uninvolved foot is assigned a reference value of 100 points. The participant then rates the involved foot on a scale ranging from 0 to 100, with higher scores indicating better self-perceived functional ability in daily life.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
score on a scale | 92.27 (6.27) | 93.73 (4.26)

13. Secondary Outcome: The Foot and Ankle Ability Measures- Sports (Self- Awareness Score)
Description: The Sports (self-awareness score) is a self-reported measure in which the participant rates the perceived functional ability of the involved (patient) foot during sports-related activities relative to the uninvolved (healthy) foot. The uninvolved foot is assigned a reference value of 100 points. The participant then rates the involved foot on a scale ranging from 0 to 100, with higher scores indicating better self-perceived sports-related functional ability.
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
score on a scale | 86.67 (5.27) | 88.13 (11.79)

14. Secondary Outcome: Y Balance- Posterolateral Direction
Description: as for outcome 7
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: % of leg length
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
% of leg length | 103.17 (6.77) | 97.19 (6.13)

15. Secondary Outcome: Y Balance- Posteromedial Direction
Description: as for outcome 7
Time Frame: Within one week after 12 treatment sessions
Measure: Mean (Standard Deviation); unit: % of leg length
Arm/Group | Exercise Group | Neurodynamic Group
Number analyzed (Participants) | 18 | 18
% of leg length | 98.13 (6.32) | 94.62 (6.35)

ADVERSE EVENTS:
Time Frame: during the experiment, up to 24 hours
Description: no any adverse event.
Arm/Group | Exercise Group | Neurodynamic Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT05090423/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT05090423/ICF_001.pdf